CLINICAL TRIAL: NCT02908425
Title: Human Metabolism of HMB
Brief Title: Cholesterol and Statin in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-0767
Record Dates: First submitted 2016-09-15; First posted 2016-09-21 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Elevated HMB Excretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy taking statin (Other): healthy subjects currently taking cholesterol lowering statin
  Interventions: Other: Statin user

INTERVENTIONS:
Other: Statin user — Subjects will be studied on 2 occasions with both being identical. One will be after 7 days or more of cholesterol lowering statin administration and the other occasion will be after at least 4 weeks of cholesterol lowering statin discontinuation. All study visits include (but are not limited to) blood draws, urine collection, and stable isotope infusions.

SUMMARY:
Statins are a class of drugs that are the most commonly prescribed medications in developing countries. Statins act on the enzyme HMG-CoA reductase to inhibit its conversion to mevalonate, a precursor for cholesterol synthesis. Subsequently statins are prescribed to patients with relatively high blood cholesterol levels. However, taking statins does not come without side effects. Most notably, the effects of statins on muscle wasting have been studied extensively. This includes up-regulation of the ubiquitin proteasome system, muscle cell damage and rhabdomyolysis, elevated creatine kinase, and mitochondrial dysfunction. Due to the negative side effects of statin therapy, additional therapies are warranted to help offset the effects on muscle wasting.

Loss of muscle mass is a significant concern as it is associated with a reduction in muscle strength and power (Ferrando et al., 1996; Creditor, 1993). This condition is observed in aging, disease states, and long periods of unloading such as hospital admission and can lead to disability, increased falls, loss of independence, and mortality. Subsequently, there is a critical need to develop interventions to counteract this loss of muscle mass and strength. Exercise is one such intervention, however, in some cases may not be a feasible option. For instance, exercise has been demonstrated to exacerbate the muscle side of effects of statins. Subjects complain of increased muscle soreness and have elevated creatine kinase levels and they also do not want to take statins anymore (Kearns et al., 2008; Parker et al., 2012; Sinzinger et al., 2004). Because of this limitation, there is a critical need to develop other interventions that can prevent the loss of muscle mass during statin use.

DETAILED DESCRIPTION:
The use of nutritional interventions have gained much attention and are being explored for their ability to increase muscle mass and/or attenuate loss of muscle mass. Leucine, isoleucine, and valine are branched chain amino acids that have been studied extensively and have been shown to stimulate muscle anabolism. Beta-hydroxy-beta-methylbutyrate (HMB), a metabolite of leucine, has been suggested to play a significant role in preserving muscle mass in situations that favor muscle mass loss. This is thought to occur through stabilizing sarcolemma integrity, reduced proteasome activity and expression of the proteasome 20S subunit, inhibition of apoptosis, and by activation of skeletal muscle satellite cells. Furthermore, in a catabolic-induced myotube and a murine adenocarcinoma cell line, HMB (50µM) was more potent in reversing the increased protein degradation and decreased protein synthesis compared to a higher dose of leucine (1mM). Similar findings were reported in a rodent cancer model. These data suggests that HMB plays a significant role in preventing muscle wasting.

Understanding the metabolic fate of HMB is crucial to developing strategies to increase HMB concentrations in populations that are subjected to muscle wasting. The objective of this application is to determine if a cholesterol lowering statin alters HMB metabolism in healthy adults. The Researchers will test the hypotheses that with statin administration, HMB metabolism and urinary excretion is affected and that this will have an unknown effect on the production of HMB and the response to intake of HMB precursors like leucine.

ELIGIBILITY:
Inclusion criteria:

* Male and Female, Age ≥ 65 y to 80 y
* BMI >20 but less than or equal to 35
* Currently taking a cholesterol lowering statin
* Stable body-weight (± 5%) for the past 3 months
* Subject is judged to be in satisfactory health based on medical history, physical examination, and laboratory screening evaluations.
* Ability to walk, sit down and stand up independently
* Ability to lie in supine or elevated position for up to 8 hours
* Willingness and ability to comply with the protocol

Exclusion criteria:

* Metabolic diseases including diabetes, hepatic or renal disorder
* Subject has malignant disease or autoimmune disease
* Subject has impaired liver function
* Subject has had a significant cardiovascular event (e.g. myocardial infarction, stroke) ≤ 6 months prior to screening visit; or stated history of congestive heart failure
* Subject has current significantly impaired liver function in the opinion of the study PI (mild asymptomatic fatty liver is acceptable), or hepatic enzyme tests are ≥2.5 times normal limit
* Subject has a chronic, contagious, infectious disease, such as active tuberculosis, hepatitis B or C, or HIV
* Subject has chronic disease such as COPD
* Subject is expected to have surgery within one-month of screening
* Subject is currently participating or has participated in a study with an investigational compound or device within 30 days of signing the informed consent.
* Presence of acute illness or metabolically unstable chronic illness (unrelated to the primary disease)
* Unwilling to stop taking nutritional protein supplements within 5 days of first study day
* Any other condition according to the PI or nurse that would interfere with the study or safety of the subject or influence the results
* Presence of fever within the last 3 days
* Untreated metabolic diseases including hepatic or renal disorder unrelated to the primary disease
* Active dependence of alcohol or drugs
* Medication: Use of substances known to influence amino acid metabolism: antibiotics within 3 weeks prior to the study visit, current use of corticosteroids, growth hormone, testosterone, estrogen, immunosuppressant, blood thinners, or insulin.
* Subject cannot refrain from taking dietary supplements/substances that could modulate metabolism or weight in the opinion of the principal investigator or physician, starting four weeks prior to enrollment and over the entire course of the study such as b-hydroxy-b-methyl butyrate (HMB) or products containing HMB
* Adherence to a weight loss diet.
* Currently taking any drugs that impact liver function
* Subject having elevated blood CK/CPK levels (3-10X above normal range)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Beta Hydroxymethyl butyrate turnover | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 minutes
  Measures the rate that Beta Hydroxymethyl butyrate is appears in blood

SECONDARY OUTCOMES:
Ketoisocapric acid turnover | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Measures the rate that Ketoisocapric acid is appears in blood
Leucine turnover | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Measures the rate that Leucine is appears in blood
Isoleucine turnover | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Measures the rate that Isoleucine is appears in blood
Ketomethylvalerate turnover | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Measures the rate that Ketomethylvalerate is appears in blood
Valine turnover | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Measures the rate that Valine is appears in blood
Ketoisovalerate turnover | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Measures the rate that Ketoisovalerate is appears in blood
Beta Hydroxymethyl butyrate concentration | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Blood Beta Hydroxymethyl butyrate concentration
Ketoisocapric acid concentration | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Blood Ketoisocapric acid concentration
Leucine concentration | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Blood Leucine concentration
Isoleucine concentration | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Blood Isoleucine concentration
Ketomethylvalerate concentration | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Blood Ketomethylvalerate concentration
Valine concentration | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Blood Valine concentration
Ketoisovalerate concentration | 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 240 min
  Blood Ketoisovalerate concentration
Beta Hydroxymethyl butyrate concentration | 0 and 240 min
  Urinary Beta Hydroxymethyl butyrate concentration

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, PHD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pallottini V. 3-Hydroxy-3-methylglutaryl-coenzyme A reductase modulator: toward age- and sex-personalized medicine. Expert Opin Ther Pat. 2015;25(10):1079-83. doi: 10.1517/13543776.2015.1061996. Epub 2015 Jul 1. PMID 26135220
- [Background] Hanai J, Cao P, Tanksale P, Imamura S, Koshimizu E, Zhao J, Kishi S, Yamashita M, Phillips PS, Sukhatme VP, Lecker SH. The muscle-specific ubiquitin ligase atrogin-1/MAFbx mediates statin-induced muscle toxicity. J Clin Invest. 2007 Dec;117(12):3940-51. doi: 10.1172/JCI32741. PMID 17992259
- [Background] Thompson PD, Clarkson P, Karas RH. Statin-associated myopathy. JAMA. 2003 Apr 2;289(13):1681-90. doi: 10.1001/jama.289.13.1681. PMID 12672737
- [Background] Phillips PS, Haas RH, Bannykh S, Hathaway S, Gray NL, Kimura BJ, Vladutiu GD, England JD; Scripps Mercy Clinical Research Center. Statin-associated myopathy with normal creatine kinase levels. Ann Intern Med. 2002 Oct 1;137(7):581-5. doi: 10.7326/0003-4819-137-7-200210010-00009. PMID 12353945
- [Background] Kaufmann P, Torok M, Zahno A, Waldhauser KM, Brecht K, Krahenbuhl S. Toxicity of statins on rat skeletal muscle mitochondria. Cell Mol Life Sci. 2006 Oct;63(19-20):2415-25. doi: 10.1007/s00018-006-6235-z. PMID 17013560
- [Background] Ferrando AA, Lane HW, Stuart CA, Davis-Street J, Wolfe RR. Prolonged bed rest decreases skeletal muscle and whole body protein synthesis. Am J Physiol. 1996 Apr;270(4 Pt 1):E627-33. doi: 10.1152/ajpendo.1996.270.4.E627. PMID 8928769
- [Background] Creditor MC. Hazards of hospitalization of the elderly. Ann Intern Med. 1993 Feb 1;118(3):219-23. doi: 10.7326/0003-4819-118-3-199302010-00011. PMID 8417639
- [Background] Kearns AK, Bilbie CL, Clarkson PM, White CM, Sewright KA, O'Fallon KS, Gadarla M, Thompson PD. The creatine kinase response to eccentric exercise with atorvastatin 10 mg or 80 mg. Atherosclerosis. 2008 Sep;200(1):121-5. doi: 10.1016/j.atherosclerosis.2007.12.029. Epub 2008 Feb 7. PMID 18261731
- [Background] Parker BA, Augeri AL, Capizzi JA, Ballard KD, Troyanos C, Baggish AL, D'Hemecourt PA, Thompson PD. Effect of statins on creatine kinase levels before and after a marathon run. Am J Cardiol. 2012 Jan 15;109(2):282-7. doi: 10.1016/j.amjcard.2011.08.045. Epub 2011 Oct 28. PMID 22036108
- [Background] Sinzinger H, O'Grady J. Professional athletes suffering from familial hypercholesterolaemia rarely tolerate statin treatment because of muscular problems. Br J Clin Pharmacol. 2004 Apr;57(4):525-8. doi: 10.1111/j.1365-2125.2003.02044.x. PMID 15025753
- [Background] Stein TP, Schluter MD, Leskiw MJ, Boden G. Attenuation of the protein wasting associated with bed rest by branched-chain amino acids. Nutrition. 1999 Sep;15(9):656-60. doi: 10.1016/s0899-9007(99)00120-3. PMID 10467608
- [Background] Stein TP, Donaldson MR, Leskiw MJ, Schluter MD, Baggett DW, Boden G. Branched-chain amino acid supplementation during bed rest: effect on recovery. J Appl Physiol (1985). 2003 Apr;94(4):1345-52. doi: 10.1152/japplphysiol.00481.2002. Epub 2002 Dec 6. PMID 12471043
- [Background] Stout JR, Smith-Ryan AE, Fukuda DH, Kendall KL, Moon JR, Hoffman JR, Wilson JM, Oliver JS, Mustad VA. Effect of calcium beta-hydroxy-beta-methylbutyrate (CaHMB) with and without resistance training in men and women 65+yrs: a randomized, double-blind pilot trial. Exp Gerontol. 2013 Nov;48(11):1303-10. doi: 10.1016/j.exger.2013.08.007. Epub 2013 Aug 24. PMID 23981904
- [Background] Deutz NE, Pereira SL, Hays NP, Oliver JS, Edens NK, Evans CM, Wolfe RR. Effect of beta-hydroxy-beta-methylbutyrate (HMB) on lean body mass during 10 days of bed rest in older adults. Clin Nutr. 2013 Oct;32(5):704-12. doi: 10.1016/j.clnu.2013.02.011. Epub 2013 Mar 4. PMID 23514626
- [Background] May PE, Barber A, D'Olimpio JT, Hourihane A, Abumrad NN. Reversal of cancer-related wasting using oral supplementation with a combination of beta-hydroxy-beta-methylbutyrate, arginine, and glutamine. Am J Surg. 2002 Apr;183(4):471-9. doi: 10.1016/s0002-9610(02)00823-1. PMID 11975938
- [Background] Nissen SL, Abumrad NN. Nutritional role of the leucine metabolite β-hydroxy β-methylbutyrate (HMB). The Journal of nutritional biochemistry. 1997;8(6):300-11.
- [Background] Smith HJ, Mukerji P, Tisdale MJ. Attenuation of proteasome-induced proteolysis in skeletal muscle by beta-hydroxy-beta-methylbutyrate in cancer-induced muscle loss. Cancer Res. 2005 Jan 1;65(1):277-83. PMID 15665304
- [Background] Hao Y, Jackson JR, Wang Y, Edens N, Pereira SL, Alway SE. beta-Hydroxy-beta-methylbutyrate reduces myonuclear apoptosis during recovery from hind limb suspension-induced muscle fiber atrophy in aged rats. Am J Physiol Regul Integr Comp Physiol. 2011 Sep;301(3):R701-15. doi: 10.1152/ajpregu.00840.2010. Epub 2011 Jun 22. PMID 21697520
- [Background] Alway SE, Pereira SL, Edens NK, Hao Y, Bennett BT. beta-Hydroxy-beta-methylbutyrate (HMB) enhances the proliferation of satellite cells in fast muscles of aged rats during recovery from disuse atrophy. Exp Gerontol. 2013 Sep;48(9):973-84. doi: 10.1016/j.exger.2013.06.005. Epub 2013 Jul 4. PMID 23832076
- [Background] Mirza KA, Pereira SL, Voss AC, Tisdale MJ. Comparison of the anticatabolic effects of leucine and Ca-beta-hydroxy-beta-methylbutyrate in experimental models of cancer cachexia. Nutrition. 2014 Jul-Aug;30(7-8):807-13. doi: 10.1016/j.nut.2013.11.012. Epub 2013 Dec 4. PMID 24984997
- [Background] Smith KL, Tisdale MJ. Increased protein degradation and decreased protein synthesis in skeletal muscle during cancer cachexia. Br J Cancer. 1993 Apr;67(4):680-5. doi: 10.1038/bjc.1993.126. PMID 8471425